CLINICAL TRIAL: NCT00946803
Title: A Patient-Controlled Cognitive-Behavioral Intervention for Cancer Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CO08316; 1R21NR010746 (NIH)
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Pain; Fatigue; Sleep Disturbance; Cancer
Keywords: Pain; Fatigue; Sleep; Cancer; Complementary therapies
MeSH Terms: conditions — Pain; Fatigue; Parasomnias; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PC-CB Intervention (Experimental): Patient-Controlled Cognitive-Behavioral Intervention
  Interventions: Behavioral: Patient-Controlled Cognitive-Behavioral Intervention
- Wait list (No Intervention): Wait list control group. Offered PC-CB Intervention after the study.

INTERVENTIONS:
Behavioral: Patient-Controlled Cognitive-Behavioral Intervention — Selection of 12 recorded imagery- and non imagery-based cognitive-behavioral coping strategies provided on an MP3 player to be used at least once per day or more frequently, as needed for pain, fatigue, and sleep disturbance.
  Arms: PC-CB Intervention

SUMMARY:
Patients receiving treatment for advanced cancer often experience co-occuring pain, fatigue, and sleep disturbance that are not relieved with medications. Brief cognitive-behavioral coping strategies such as relaxation or imagery have been shown to be useful for these symptoms individually and may be effective for the cluster of co-occuring pain, fatigue, and sleep disturbance. Because single cognitive-behavioral strategies don't work equally well for all persons, providing training in multiple cognitive-behavioral strategies is necessary. However, oncology nurses report having insufficient time and are often not available to deliver the interventions exactly when patients experience symptom exacerbation. This application proposes a patient-controlled cognitive-behavioral (PC-CB) intervention, using an MP3 player to deliver recorded cognitive-behavioral strategies. The PC-CB intervention would allow patients to select from a variety of cognitive-behavioral strategies based on their personal preferences, and facilitate self-administration of those strategies at whatever time and place the symptoms occur, without increasing burden on nursing staff. Primary aims are (1) to explore acceptability and patterns of use of the recorded cognitive-behavioral strategies and (2) to pilot test efficacy of the PC-CB intervention compared to a waitlist control.

DETAILED DESCRIPTION:
Patients undergoing treatment for advanced cancer often experience the combination of pain, fatigue, and sleep disturbance as symptoms that co-occur or "cluster" within patients. Medications may be effective in reducing some of these symptoms; however, they often have side effects that exacerbate the other symptoms. Practice guidelines and research evidence suggest that cognitive-behavioral (CB) strategies may be effective treatments with few, if any, side effects for each of these symptoms. However, investigators have not yet explored the effect of CB strategies on co-occuring pain, fatigue, and sleep disturbance. It is possible that an intervention that is effective for one symptom may also have beneficial effects on the other co-occuring symptoms. For example, controlling pain may permit better sleep and subsequently reduce fatigue. Cognitive-behavioral strategies, however, are not equally effective for all patients, and training in just one strategy may not be sufficient. Providing multiple CB strategies may be more efficacious, but is complicated by the fact that oncology nurses report having insufficient time and equipment to deliver the interventions in practice. And given patient-care demands, providing CB strategies exactly when patients experience increased symptom intensity is usually not feasible. A patient-centered approach to symptom management would allow patients to select from a variety of CB strategies based on their personal preferences, skills, and interests and permit the use of those strategies at whatever time and place the symptoms occur. The use of MP3 technology to deliver the intervention would allow patients to control delivery of the CB strategies without increasing burden on nursing staff and could potentially improve all symptoms in the cluster. The purpose of this study is to conduct a pilot test of a 2-week patient-controlled cognitive-behavioral intervention (PC-CB intervention), using an MP3 player to deliver recorded CB strategies for co-occurring pain, fatigue, and sleep disturbance during cancer treatment.

Primary Aims

1. To explore the acceptability and patterns of use of recorded CB strategies delivered via MP3 player among patients receiving treatment for advanced cancer.
2. To pilot test efficacy of a 2-week PC-CB intervention on symptom outcomes during cancer treatment compared to a waitlist control condition.

Secondary Aims

1. To determine if changes in perceived control over symptoms and outcome expectancy mediate the effect of the PC-CB intervention on symptom outcomes.
2. To determine if gender, age, imaging ability, and concurrent symptoms moderate the impact of the PC-CB intervention on symptom outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Advanced (metastatic/recurrent) lung, prostate, colorectal, or GYN cancer.
* Currently receiving chemotherapy or radiation treatments.
* Worst pain, fatigue, sleep disturbance rated 3 or greater on 0 - 10 scale.

Exclusion Criteria:

* Pain that is post-operative (< 3 months since surgery) or neuropathic in etiology.
* Hospitalized for psychiatric reasons within the last 3 months.
* Unable to read, write, or understand English.
* Diagnosis of confusion or cognitive impairment that would preclude completion of study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
symptom severity | two weeks

SECONDARY OUTCOMES:
symptom interference with daily activities | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Kwekkeboom, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Kwekkeboom KL, Abbott-Anderson K, Cherwin C, Roiland R, Serlin RC, Ward SE. Pilot randomized controlled trial of a patient-controlled cognitive-behavioral intervention for the pain, fatigue, and sleep disturbance symptom cluster in cancer. J Pain Symptom Manage. 2012 Dec;44(6):810-22. doi: 10.1016/j.jpainsymman.2011.12.281. Epub 2012 Jul 7. PMID 22771125